CLINICAL TRIAL: NCT05736731
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of A2B530, an Autologous Logic-gated Tmod™ Chimeric Antigen Receptor T Cell (CAR T), in Heterozygous HLA-A*02 Adult Subjects With Recurrent Unresectable, Locally Advanced, or Metastatic Solid Tumors That Express CEA and Have Lost HLA-A*02 Expression
Brief Title: A Study to Evaluate the Safety and Efficacy of A2B530, a Logic-gated CAR T, in Participants With Solid Tumors That Express CEA and Have Lost HLA-A*02 Expression
Acronym: EVEREST-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: A2 Biotherapeutics Inc. (Industry)
Collaborators: Tempus AI (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2B530-101
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor, Adult; Solid Tumor; Pancreatic Cancer; Pancreatic Neoplasms; Pancreas Cancer; Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Recurrent; Non-Small Cell Squamous Lung Cancer; NSCLC; NSCLC, Recurrent; Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenocarcinoma; CRC; Colorectal Cancer Metastatic; Cancer
Keywords: CAR T Cell; Solid Tumors; autologous; T cell; Carcinoembryonic Antigen; CEA; HLA-A2; Solid Tumors Expressing CEA; Pancreatic Cancer; PANC; CRC; Colorectal Cancer; NSCLC; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Recurrence; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- A2530 (Experimental): Patients receive Preconditioning Lymphodepletion (PCLD) Regimen followed by a single dose of A2B530 intravenously on day 0
  Interventions: Biological: A2B530; Diagnostic Test: xT-Onco with HLA-LOH Assay

INTERVENTIONS:
Biological: A2B530 — Autologous logic-gated Tmod CAR T-cells
  Other Names: Tmod CAR T-cell Therapy
Diagnostic Test: xT-Onco with HLA-LOH Assay — An investigational next generation sequencing (NGS) in vitro diagnostic (IVD) medical device

SUMMARY:
The goal of this study is to test A2B530,an autologous logic-gated Tmod™ CAR T-cell product in subjects with solid tumors including colorectal cancer (CRC), pancreatic cancer (PANC), non-small cell lung cancer (NSCLC), and other solid tumors that express CEA and have lost HLA-A*02 expression.

The main questions this study aims to answer are:

* Phase 1: What is the maximum or recommended dose of A2B530 that is safe for patients
* Phase 2: Does the recommended dose of A2B530 kill the solid tumor cells and protect the patient's healthy cells

Participants will be required to perform study procedures and assessments, and will also receive the following study treatments:

* Enrollment and Apheresis in BASECAMP-1 (NCT04981119)
* Preconditioning Lymphodepletion (PCLD) Regimen
* A2B530 Tmod CAR T cells at the assigned dose

DETAILED DESCRIPTION:
This is a phase 1/2, multi-center, open-label study that enrolls adult subjects with recurrent unresectable, locally advanced, or metastatic (considered non-curative) CRC, NSCLC, PANC, or other solid tumors with CEA expression. Subjects must be germline HLA-A*02 heterozygous, with tumors that express CEA and somatic loss of HLA-A*02. The purpose of Phase 1 of this study is to determine the safety and the optimal dose of A2B530 (after PCLD) in participants with solid tumor disease. The purpose of Phase 2 of this study is to determine the further safety and efficacy (how well it treats the solid tumor disease) of A2B530.

The treatment available for these cancers and other solid tumors can be toxic, debilitating, and fatal. In the recurrent unresectable, locally advanced, or metastatic setting, the intent of standard of care treatment is typically palliative rather than curative, and has not changed significantly in several decades. A2 Bio hypothesizes that A2B530 Tmod CAR T-cell therapy will enable the killing of tumor target cells (those cells that express CEA and have LOH for HLA-A*02 protein). Additionally, normal healthy cells that maintain HLA-A*02 expression and co-express CEA (eg, gut mucosal tissue) will not be targeted due to the blocker portion of the Tmod CAR T cell that acts as a self-regulated safety switch that protects normal tissue from damage. A2 Bio believes this will provide a therapeutic safety window compared to previous solid tumor targeting therapies. This hypothesis will be explored in the study.

Participants for this study must enroll and have their T cells collected (apheresis) in the pre-screening BASECAMP-1 study (NCT04981119). T cells are collected, processed and stored for each participant. Upon disease progression the participant may screen for this study (EVEREST-1) and the participant's T cells are then manufactured and infused following PCLD regimen. There is no time requirement between the studies, and patients may go directly from BASECAMP-1 to EVEREST-1 based on their own disease course.

ELIGIBILITY:
Key Inclusion Criteria:

1. Appropriately enrolled in the BASECAMP-1 A2 Biotherapeutics, Inc. study, with tissue demonstrating LOH of HLA-A*02:01 by NGS (whenever possible from the primary site), successful apheresis and PBMC processing, and with sufficient stored cells available for Tmod CAR T-cell therapy
2. Histologically confirmed recurrent unresectable, locally advanced, or metastatic CRC, NSCLC, PANC, or other solid tumors associated with CEA expression. Measurable disease is required with lesions of >1.0 cm by computed tomography (CT). (Soluble CEA is not acceptable as the sole measure of disease).
3. Received previous required therapy for the appropriate solid tumor disease as described in the protocol
4. Has adequate organ function as described in the protocol
5. ECOG performance status of 0 to 1
6. Life expectancy of ≥3 months
7. Willing to comply with study schedule of assessments including long term safety follow up

Key Exclusion Criteria:

1. Has disease that is suitable for local therapy or able to receive standard of care therapy that is therapeutic and not palliative
2. Prior allogeneic stem cell transplant
3. Prior solid organ transplant
4. Cancer therapy within 3 weeks or 3 half lives of A2B530 infusion
5. Radiotherapy within 28 days of A2B530 infusion
6. Unstable angina, arrhythmia, myocardial infarction, or any other significant cardiac disease within the last 6 months
7. Any new symptomatic pulmonary embolism (PE) or a deep vein thrombosis (DVT) within 3 months of enrollment. Therapeutic dosing of anticoagulants is allowed for history of PE or DVT if greater than 3 months from time of enrollment, and adequately treated.
8. Requires supplemental home oxygen
9. Females of childbearing potential who are pregnant or breastfeeding
10. Subjects, both male and female, of childbearing potential who are not willing to practice birth control from the time of consent through 6 months post infusion of A2B530

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Rate of adverse events and dose limiting toxicities (DLTs) by dose level | From the time of Informed consent until 24 months (2 years) post A2B530 infusion.
  Adverse Events and toxicity will be evaluated according to the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version 5.0 (or current version). Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) events will be graded according to the criteria described in the current protocol.
Phase 1: Recommended Phase 2 Dose (RP2D) | 21 days post A2B530 infusion
  The RP2D will be identified utilizing a BOIN study design in addition to considering safety and biomarker analysis.
Phase 2: The Overall Response Rate (ORR) for patients | 24 months post A2B530 infusion
  The ORR will be evaluated per RECIST v1.1 and assessed by independent central review.

SECONDARY OUTCOMES:
Persistence of A2B530 | up to 24 months post A2B530 infusion
  Number of A2B530 Tmod CAR T cells present in patients treated with A2B530 as assessed by Polymerase Chain Reaction (PCR) (or similar method) on participant blood samples
Cytokine analysis | up to 24 months post A2B530 infusion
  Cytokine levels in patients treated with A2B530 assessed by cytokine analysis on participant blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ng, MD, Study Director — A2 Biotherapeutics Inc.
Locations (8):
- United States (8):
  - Banner Health, Gilbert, Arizona
  - University of California San Diego, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared within 1 year of study completion.
Supporting Information: CSR
Time Frame: Data will be available within 1 year of the completion of the study, the length of time of availability is to be determined.

REFERENCES:
- [Background] Hamburger AE, DiAndreth B, Cui J, Daris ME, Munguia ML, Deshmukh K, Mock JY, Asuelime GE, Lim ED, Kreke MR, Tokatlian T, Kamb A. Engineered T cells directed at tumors with defined allelic loss. Mol Immunol. 2020 Dec;128:298-310. doi: 10.1016/j.molimm.2020.09.012. Epub 2020 Oct 1. PMID 33012527
- [Background] Hwang MS, Mog BJ, Douglass J, Pearlman AH, Hsiue EH, Paul S, DiNapoli SR, Konig MF, Pardoll DM, Gabelli SB, Bettegowda C, Papadopoulos N, Vogelstein B, Zhou S, Kinzler KW. Targeting loss of heterozygosity for cancer-specific immunotherapy. Proc Natl Acad Sci U S A. 2021 Mar 23;118(12):e2022410118. doi: 10.1073/pnas.2022410118. PMID 33731480
- [Background] Perera J, Mapes B, Lau D, et al. Detection of human leukocyte antigen class I loss of heterozygosity in solid tumor types by next-generation DNA sequencing. J Immunother Cancer. 2019, 7(Suppl 1):P103
- [Background] Beroukhim R, Mermel CH, Porter D, Wei G, Raychaudhuri S, Donovan J, Barretina J, Boehm JS, Dobson J, Urashima M, Mc Henry KT, Pinchback RM, Ligon AH, Cho YJ, Haery L, Greulich H, Reich M, Winckler W, Lawrence MS, Weir BA, Tanaka KE, Chiang DY, Bass AJ, Loo A, Hoffman C, Prensner J, Liefeld T, Gao Q, Yecies D, Signoretti S, Maher E, Kaye FJ, Sasaki H, Tepper JE, Fletcher JA, Tabernero J, Baselga J, Tsao MS, Demichelis F, Rubin MA, Janne PA, Daly MJ, Nucera C, Levine RL, Ebert BL, Gabriel S, Rustgi AK, Antonescu CR, Ladanyi M, Letai A, Garraway LA, Loda M, Beer DG, True LD, Okamoto A, Pomeroy SL, Singer S, Golub TR, Lander ES, Getz G, Sellers WR, Meyerson M. The landscape of somatic copy-number alteration across human cancers. Nature. 2010 Feb 18;463(7283):899-905. doi: 10.1038/nature08822. PMID 20164920
- [Background] Sandberg ML, Wang X, Martin AD, Nampe DP, Gabrelow GB, Li CZ, McElvain ME, Lee WH, Shafaattalab S, Martire S, Fisher FA, Ando Y, Liu E, Ju D, Wong LM, Xu H, Kamb A. A carcinoembryonic antigen-specific cell therapy selectively targets tumor cells with HLA loss of heterozygosity in vitro and in vivo. Sci Transl Med. 2022 Mar 2;14(634):eabm0306. doi: 10.1126/scitranslmed.abm0306. Epub 2022 Mar 2. PMID 35235342
- See also: A2 Biotherapeutics Inc. — http://www.a2bio.com
- See also: BASECAMP-1 Study — https://clinicaltrials.gov/ct2/show/NCT04981119?term=LOH+Apheresis&cond=Cancer&cntry=US&draw=2&rank=1